CLINICAL TRIAL: NCT03844789
Title: The International Diabetes Closed Loop (iDCL) Trial: Clinical Acceptance of the Artificial Pancreas in Pediatrics: A Study of t:Slim X2 With Control-IQ Technology
Brief Title: A Study of t:Slim X2 With Control-IQ Technology
Acronym: DCLP5
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: Tandem Diabetes Care, Inc. (Industry); DexCom, Inc. (Industry); Jaeb Center for Health Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: DCLP5
Record Dates: First submitted 2019-02-14; First posted 2019-02-18 (Actual); Results first posted 2023-04-10 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-03

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Artificial Pancreas (AP); Control-IQ System; Insulin Pump; Closed Loop Control (CLC); Continuous Glucose Monitor (CGM); Multiple Daily Injections (MDI); Sensor Augmented Pump (SAP)
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Closed Loop Control (CLC) (Experimental): Eligible participants not currently using an insulin pump and Dexcom G4, G5 or Dexcom G6 CGM with minimum data requirements will initiate a run-in phase of 2 to 4 weeks that will be customized based on whether the participant is already a pump or CGM user. Participants who skip or successfully complete the run-in will be randomly assigned 3:1 to the use of closed-loop control (CLC group) system using Tandem Control-IQ Technology & Dexcom G6 CGM vs Control Group for 16 weeks. Participants randomized to the closed loop control (CLC) arm will use the t:slim X2 with Control-IQ Technology & Dexcom G6 CGM for 16 weeks. All participants will be provided the option of continue using the t:slim X2 with Control-IQ system in a 12 week Extension Phase.
  Interventions: Device: t:slim X2 with Control-IQ Technology & Dexcom G6 CGM
- Control Group (Active Comparator): Eligible participants not currently using an insulin pump and Dexcom G4, G5 or Dexcom G6 CGM with minimum data requirements will initiate a run-in phase of 2 to 4 weeks that will be customized based on whether the participant is already a pump or CGM user. Participants who skip or successfully complete the run-in will be randomly assigned 3:1 to the use of closed-loop control (CLC group) system using Tandem t:slim X2 with Control-IQ Technology vs Control Group for 16 weeks. All participants will be provided the option of using t:slim X2 with Control-IQ system in a 12 week Extension Phase.
  Interventions: Device: Control Group

INTERVENTIONS:
Device: t:slim X2 with Control-IQ Technology & Dexcom G6 CGM — Eligible participants will be use the t:slim X2 with Control-IQ Technology & Dexcom G6 CGM technology for 16 weeks during the main study. All participants will be provided the option of continue using the t:slim X2 with Control-IQ system in a 12 week Extension Phase. This arm to be uset:slim X2 with Control-IQ Technology & Dexcom G6 CGM
  Other Names: Experimental
  Arms: Closed Loop Control (CLC)
Device: Control Group — Eligible participants will be use the study Dexcom G6 CGM for 16 weeks during the main study. All participants will be provided the option of using the t:slim X2 with Control-IQ system in a 12 week Extension Phase.
  Other Names: Sensor-Augmented Pump (SAP)
  Arms: Control Group

SUMMARY:
The purpose of this study is to learn whether an investigational automated insulin delivery system ("study system") for children with type 1 diabetes can safely improve blood glucose (sometimes called blood sugar) control. The system uses continuous glucose monitoring (CGM), an insulin pump, and a software algorithm to automatically give insulin and control blood glucose. This is called a "closed-loop control" system.

DETAILED DESCRIPTION:
After consent is signed, eligibility will be assessed. Eligible participants not currently using an insulin pump and Dexcom CGM with minimum data requirements will initiate a run-in phase of 2-4 weeks that will be customized based on whether the participant is already a pump or CGM user. Participants who skip or successfully complete the run-in will be randomly assigned 3:1 to the use of closed-loop control (CLC group) using t:slim X2 with Control-IQ Technology vs. Control Group for 16 weeks. The Control Group will be offered to transition to use CLC and the experimental arm will extend their use of CLC for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis, based on investigator assessment, of type 1 diabetes for at least one year and using insulin for at least 6 months
2. Familiarity and use of a carbohydrate ratio for meal boluses.
3. Age ≥ 6 and ≤ 13 years old
4. Weight ≥25 kg and ≤140 kg
5. For females, not currently known to be pregnant If female and sexually active, must agree to use a form of contraception to prevent pregnancy while a participant in the study. A negative serum or urine pregnancy test will be required for all females of child-bearing potential. Participants who become pregnant will be discontinued from the study. Also, participants who during the study develop and express the intention to become pregnant within the timespan of the study will be discontinued.
6. Living with one or more parent/legal guardian knowledgeable about emergency procedures for severe hypoglycemia and able to contact emergency services and study staff.
7. Willingness to suspend use of any personal closed loop system that they use at home for the duration of the clinical trial once the study CGM is in use
8. Investigator has confidence that the participant can successfully operate all study devices and is capable of adhering to the protocol
9. Willingness to switch to lispro (Humalog) or aspart (Novolog) if not using already, and to use no other insulin besides lispro (Humalog) or aspart (Novolog) during the study for participants using to t:slim X2. This includes:

   * Participants randomized to Control IQ
   * Participants on the SAP group on MDI treatment that will be provided a Tandem pump to switch to CSII
   * Participates that are already in Continuous Subcutaneous Insulin Infusion (CSII) randomized to SAP during the extension phase when transition to Control IQ
10. Total daily insulin dose (TDD) at least 10 U/day
11. Willingness not to start any new non-insulin glucose-lowering agent during the course of the trial
12. Participant and parent(s)/guardian(s) willingness to participate in all training sessions as directed by study staff.

Exclusion Criteria:

1. Concurrent use of any non-insulin glucose-lowering agent other than metformin (including glucagon-like peptide [GLP-1] agonists, Symlin, dipeptidyl peptidase 4 [DPP-4] inhibitors, sodium-glucose cotransporter-2 (SGLT2) inhibitors, sulfonylureas).
2. Hemophilia or any other bleeding disorder
3. A condition, which in the opinion of the investigator or designee, would put the participant or study at risk (specified on the study procedure manual)
4. Participation in another pharmaceutical or device trial at the time of enrollment or during the study
5. Employed by, or having immediate family members employed by Tandem Diabetes Care, Inc., or having a direct supervisor at place of employment who is also directly involved in conducting the clinical trial (as a study investigator, coordinator, etc.); or having a first-degree relative who is directly involved in conducting the clinical trial

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 101 (Actual)
Dates: Start 2019-06-06 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2020-03-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa J Schoelwer, MD, Principal Investigator — University of Virginia
Locations (4):
- United States (4):
  - Stanford University, Stanford, California
  - Barbara Davis Center, University of Colorado, Aurora, Colorado
  - Yale University, New Haven, Connecticut
  - UVA Center for Diabetes Technology, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Will follow the NIH Data Sharing Policy and Implementation Guidance on sharing research resources for research purposes to qualified individuals within the scientific community.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Generally, data will be made available after the primary publications of each study.
Access Criteria: The Data Sharing Agreements will be formulated by the Steering Committee in collaboration with the NIH Project Scientist Program Official.
  In addition, under special arrangements, complete data sets will be provided to industry partners who would use the data for regulatory clearance (PMA - pre-market approval) of the tested artificial pancreas system. This will be done in response to the specific requirements of RFA-DK-14-024 for this project to "…generate data able to satisfy safety and efficacy requirements by regulatory agencies regarding the clinical testing of artificial pancreas device systems" in the target population of people with type 1 diabetes.

REFERENCES:
- [Result] Breton MD, Kanapka LG, Beck RW, Ekhlaspour L, Forlenza GP, Cengiz E, Schoelwer M, Ruedy KJ, Jost E, Carria L, Emory E, Hsu LJ, Oliveri M, Kollman CC, Dokken BB, Weinzimer SA, DeBoer MD, Buckingham BA, Chernavvsky D, Wadwa RP; iDCL Trial Research Group. A Randomized Trial of Closed-Loop Control in Children with Type 1 Diabetes. N Engl J Med. 2020 Aug 27;383(9):836-845. doi: 10.1056/NEJMoa2004736. PMID 32846062
- [Result] Kanapka LG, Wadwa RP, Breton MD, Ruedy KJ, Ekhlaspour L, Forlenza GP, Cengiz E, Schoelwer MJ, Jost E, Carria L, Emory E, Hsu LJ, Weinzimer SA, DeBoer MD, Buckingham BA, Oliveri M, Kollman C, Dokken BB, Chernavvsky D, Beck RW; iDCL Trial Research Group. Extended Use of the Control-IQ Closed-Loop Control System in Children With Type 1 Diabetes. Diabetes Care. 2021 Feb;44(2):473-478. doi: 10.2337/dc20-1729. Epub 2020 Dec 21. PMID 33355258
- [Result] Schoelwer MJ, Kanapka LG, Wadwa RP, Breton MD, Ruedy KJ, Ekhlaspour L, Forlenza GP, Cobry EC, Messer LH, Cengiz E, Jost E, Carria L, Emory E, Hsu LJ, Weinzimer SA, Buckingham BA, Lal RA, Oliveri MC, Kollman CC, Dokken BB, Chernavvsky DR, Beck RW, DeBoer MD; iDCL Trial Research Group. Predictors of Time-in-Range (70-180 mg/dL) Achieved Using a Closed-Loop Control System. Diabetes Technol Ther. 2021 Jul;23(7):475-481. doi: 10.1089/dia.2020.0646. Epub 2021 Mar 9. PMID 33689454
- [Derived] Beck RW, Kanapka LG, Breton MD, Brown SA, Wadwa RP, Buckingham BA, Kollman C, Kovatchev B. A Meta-Analysis of Randomized Trial Outcomes for the t:slim X2 Insulin Pump with Control-IQ Technology in Youth and Adults from Age 2 to 72. Diabetes Technol Ther. 2023 May;25(5):329-342. doi: 10.1089/dia.2022.0558. Epub 2023 Apr 12. PMID 37067353
- [Derived] Cobry EC, Bisio A, Wadwa RP, Breton MD. Improvements in Parental Sleep, Fear of Hypoglycemia, and Diabetes Distress With Use of an Advanced Hybrid Closed-Loop System. Diabetes Care. 2022 May 1;45(5):1292-1295. doi: 10.2337/dc21-1778. PMID 35202468
- [Derived] Schoelwer MJ, Bisio A, Breton MD, DeBoer MD. Assessment for Predictors of Rise in Hemoglobin A1c During Extended Use of a Closed-Loop Control System. Diabetes Technol Ther. 2022 Apr;24(4):285-288. doi: 10.1089/dia.2021.0405. PMID 34962164
- [Derived] Cobry EC, Kanapka LG, Cengiz E, Carria L, Ekhlaspour L, Buckingham BA, Hood KK, Hsu LJ, Messer LH, Schoelwer MJ, Emory E, Ruedy KJ, Beck RW, Wadwa RP, Gonder-Frederick L; iDCL Trial Research Group. Health-Related Quality of Life and Treatment Satisfaction in Parents and Children with Type 1 Diabetes Using Closed-Loop Control. Diabetes Technol Ther. 2021 Jun;23(6):401-409. doi: 10.1089/dia.2020.0532. Epub 2021 Jan 28. PMID 33404325

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between June 21, 2019, and August 30, 2019, a total of 101 patients (19 to 28 per trial site) were randomly assigned to the closed-loop group (78 patients) or the control group (23 patients).
Groups:
- Closed Loop Control (CLC): Eligible participants not currently using an insulin pump and Dexcom G4, G5 or Dexcom G6 CGM with minimum data requirements will initiate a run-in phase of 2 to 4 weeks that will be customized based on whether the participant is already a pump or CGM user. Participants who skip or successfully complete the run-in will be randomly assigned 3:1 to the use of closed-loop control (CLC group) system using Tandem Control-IQ Technology & Dexcom G6 CGM vs Control Group for 16 weeks. Participants randomized to the closed loop control (CLC) arm will use the t:slim X2 with Control-IQ Technology & Dexcom G6 CGM for 16 weeks. All participants will be provided the option of continue using the t:slim X2 with Control-IQ system in a 12 week Extension Phase.
  t:slim X2 with Control-IQ Technology & Dexcom G6 CGM: Eligible participants will be use the t:slim X2 with Control-IQ Technology & Dexcom G6 CGM technology for 16 weeks during the main study. All participants will be provided the option of continue using the t:slim X2 with Control-IQ system in a 12 week Extension Phase. This arm to be use t:slim X2 with Control-IQ Technology & Dexcom G6 CGM.
Period: Main Study
Arm/Group | Closed Loop Control (CLC) | Control Group
Started | 78 | 23
16 Week Main Study | 78 | 22
Completed | 78 | 22
Not Completed | 0 | 1
Period: Extension Study
Arm/Group | Closed Loop Control (CLC) | Control Group
Started | 78 | 22
Completed | 78 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Standard of Care: Eligible participants not currently using an insulin pump and Dexcom G4, G5 or Dexcom G6 CGM with minimum data requirements will initiate a run-in phase of 2 to 4 weeks that will be customized based on whether the participant is already a pump or CGM user. Participants who skip or successfully complete the run-in will be randomly assigned 3:1 to the use of closed-loop control (CLC group) system using Tandem t:slim X2 with Control-IQ Technology vs Control Group for 16 weeks. All participants will be provided the option of using t:slim X2 with Control-IQ system in a 12 week Extension Phase.
  Control Group: Eligible participants will be use the study Dexcom G6 CGM for 16 weeks during the main study. All participants will be provided the option of using the t:slim X2 with Control-IQ system in a 12 week Extension Phase.
- Total: Total of all reporting groups
Arm/Group | Closed Loop Control (CLC) | Standard of Care | Total
Number analyzed (Participants) | 78 | 23 | 101
Age, Customized [Count of Participants; unit: Participants]
  Ages 6 to 9 | 21 | 8 | 29
  Ages 10 to 13 | 57 | 15 | 72
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 12 | 50
  Male | 40 | 11 | 51
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White, non-Hispanic | 64 | 18 | 82
  HIspanic or Latino | 6 | 2 | 8
  Black/African-American | 0 | 0 | 0
  Asian | 1 | 1 | 2
  More than one race | 7 | 2 | 9
Diabetes Duration [Count of Participants; unit: Participants] — Length of time in years since participants had been diagnosed with type I diabetes prior to screening
  Participants
    1 to 4 years | 42 | 7 | 49
    5 to 10 years | 28 | 14 | 42
    More than 10 years | 8 | 2 | 10
Insulin Modality [Count of Participants; unit: Participants]
  Insulin Pump | 62 | 19 | 81
  Multiple Daily Injection (MDI) | 16 | 4 | 20
Prior Continuous Glucose Monitor Use [Count of Participants; unit: Participants]
  Never | 2 | 0 | 2
  In past, but not current | 4 | 2 | 6
  Current | 72 | 21 | 93
Body Mass Index (BMI) Z-score [Mean (Standard Deviation); unit: Z-score] — A Z-score of zero represents the US population mean for their age group. Positive Z scores indicate higher body mass index values than the population mean, which is generally considered undesirable.
  Z-score | 0.4 (1.0) | 0.5 (1.0) | 0.45 (1.0)
Parents Education [Count of Participants; unit: Participants]
  ≤H.S. Diploma | 2 | 0 | 2
  Associates Degree or Some College but no Degree | 5 | 1 | 6
  Bachelor's Degree | 32 | 9 | 41
  Master's Degree | 34 | 11 | 45
  Doctoral or Prof Degree | 5 | 2 | 7
Annual Household Income [Count of Participants; unit: Participants]
  <$25,000 | 0 | 0 | 0
  $25,000 - <$35,000 | 2 | 0 | 2
  $35,000 - <$50,000 | 1 | 2 | 3
  $50,000 - <$75,000 | 5 | 0 | 5
  $75,000 - <$100,000 | 13 | 4 | 17
  $100,000 - <$200,000 | 27 | 8 | 35
  ≥$200,000 | 26 | 7 | 33
  Missing Data | 4 | 2 | 6
Health Insurance [Count of Participants; unit: Participants]
  Private | 70 | 21 | 91
  CHP or other government sponsored/Medicaid | 6 | 1 | 7
  Military | 2 | 1 | 3
  Other | 0 | 0 | 0
  None | 0 | 0 | 0
HbA1c Local Lab at Screening [Count of Participants; unit: Participants]
  <8.0% | 50 | 12 | 62
  8.0%<9.0% | 18 | 8 | 26
  ≥9.0% | 10 | 3 | 13
HbA1c Central Lab at Randomization [Count of Participants; unit: Participants]
  <8.0% | 50 | 11 | 61
  8.0%<9.0% | 20 | 10 | 30
  ≥9.0% | 8 | 2 | 10
Total Daily Insulin [Mean (Standard Deviation); unit: Units of Insulin per kg per day] | 0.89 (0.24) | 0.94 (0.24) | 0.92 (0.24)
C-peptide (nmol/L) [Count of Participants; unit: Participants]
  <0.2 nmol/L | 72 | 21 | 93
  ≥0.2 nmol/L | 6 | 2 | 8
Diabetic Ketoacidosis (DKA) in Last 12 Months [Count of Participants; unit: Participants] — Hyperglycemic events are classified as DKA if the following are present: Symptoms such as polyuria, polydipsia, nausea, or vomiting; Serum ketones greater than or equal to 1.5 mmol/L or large/moderate urine ketones; Either arterial blood pH <7.3 or venous pH < 7.24 or serum bicarbonate < 15; and treatment provided in a health care facility.
  Participants
    No DKA events in the last 12 months | 74 | 23 | 97
    1 DKA event in the last 12 months | 3 | 0 | 3
    2 DKA events in the last 12 months | 1 | 0 | 1
Severe Hypoglycemia (SH) in Last 12 Months [Count of Participants; unit: Participants] | 78 | 23 | 101

OUTCOME MEASURES:

1. Primary Outcome: Continuous Glucose Monitor (CGM)-Measured Percent Time in Range 70-180mg/dL Over 16 Week Trial Period
Description: The primary outcome for the first phase is percent of time participants spent in blood sugar target range 70-180 mg/dL as measured by CGM in Closed Loop Control (CLC) group vs. Control Group. Larger percentages of time spent in this range is considered to be a desirable outcome.
Time Frame: From randomization to data collection completion at the end of 16 weeks
Population: One participant in the control group was missing follow-up data.
Measure: Mean (Standard Deviation); unit: Percentage of Time
Arm/Group | Closed Loop Control (CLC) | Control Group
Number analyzed (Participants) | 78 | 22
Percentage of Time | 67 (10) | 55 (13)

2. Secondary Outcome: CGM-Measured Percent of Time Above 180 mg/dL Over 16 Week Trial Period
Description: Continuous Blood Glucose Monitor (CGM) values are generated every 5 minutes over the course of the study. Smaller percentages of CGM-measured time above 180 mg/dL is considered a positive outcome.
Time Frame: From randomization to data collection completion at the end of 16 weeks
Measure: Mean (Standard Deviation); unit: Percentage of Time
Arm/Group | Closed Loop Control (CLC) | Control Group
Number analyzed (Participants) | 78 | 22
Percentage of Time | 31 (10) | 43 (14)

3. Secondary Outcome: CGM-Measured Mean Glucose Over 16 Week Trial Period
Description: Continuous Blood Glucose Monitor (CGM) values are generated every 5 minutes over the course of the study. CGM metrics were calculated by pooling all CGM readings in the 16-week period starting from the randomization visit up through the 16 week visit. If a participant dropped out before completing the 16-week visit, all available data through the last visit date was included for calculating CGM metrics. Minimum 168 hours of CGM data was required to calculate CGM metrics. Lower mean glucose numbers as measured by CGM in mg/dL is considered a positive outcome.
Time Frame: From randomization to data collection completion at the end of 16 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Closed Loop Control (CLC) | Control Group
Number analyzed (Participants) | 78 | 22
mg/dL | 162 (18) | 179 (26)

4. Secondary Outcome: Glycated Hemoglobin A1C (HbA1c) Percent at End Of 16 Week Trial Period
Description: Glycated Hemoglobin A1C (HbA1c) is a physiological marker of the percentage of red blood cells that have glycated (bonded with a sugar). HbA1c is used to measure changes in average blood sugar over the past three months. 5-6% is normal, 7% and above is correlated with negative long-term health outcomes.
Time Frame: At data collection completion at the end of 16 weeks
Measure: Mean (Standard Deviation); unit: Percent of Hemoglobin that was Glycated
Arm/Group | Closed Loop Control (CLC) | Control Group
Number analyzed (Participants) | 78 | 22
Percent of Hemoglobin that was Glycated | 7.0 (0.8) | 7.6 (0.9)

5. Secondary Outcome: CGM-measured Percent of Time Below 70 mg/dL Over 16 Week Trial Period
Description: Continuous Blood Glucose Monitor (CGM) values are generated every 5 minutes over the course of the study. CGM measured blood sugar values below 70 mg/dL are considered to be somewhat dangerous due to the possibility of unconsciousness and death at low blood sugar values. Thus, less time spent below 70mg/dL is considered a positive outcome.
Time Frame: From randomization to data collection completion at the end of 16 weeks
Measure: Median (Inter-Quartile Range); unit: Percentage of Time
Arm/Group | Closed Loop Control (CLC) | Control Group
Number analyzed (Participants) | 78 | 22
Percentage of Time | 1.57 [0.79 to 2.44] | 1.80 [1.13 to 3.04]

6. Secondary Outcome: CGM-measured Median and Interquartile Range of Percent of Time Below 54 mg/dL Over 16 Week Trial Period
Description: GM measured blood sugar values below 54 mg/dL have the potential to lead to unconsciousness or death. Thus, less time below 54 mg/dL is considered a better outcome.
Time Frame: From randomization to data collection completion at the end of 16 weeks
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Closed Loop Control (CLC) | Control Group
Number analyzed (Participants) | 78 | 22
percentage of time | 0.23 [0.10 to 0.45] | 0.29 [0.12 to 0.62]

7. Secondary Outcome: CGM-measured Percent of Time Above 250 mg/dL Over 16 Week Trial Period
Description: CGM measured blood sugar values above 250 mg/dL are considered to be undesirable. Thus, less time spent above 250mg/dL is considered a positive outcome.
Time Frame: From randomization to data collection completion at the end of 16 weeks
Measure: Median (Inter-Quartile Range); unit: Percentage of Time
Arm/Group | Closed Loop Control (CLC) | Control Group
Number analyzed (Participants) | 78 | 22
Percentage of Time | 7.8 [5.1 to 14.3] | 18.4 [9.4 to 24.6]

8. Secondary Outcome: Continuous Glucose Monitor (CGM)-Measured Glucose Variability Measured With the Coefficient of Variation (CV) Over 16 Week Trial Period
Description: Continuous Blood Glucose Monitor (CGM) values are generated every 5 minutes over the course of the study. CGM metrics were calculated by pooling all CGM readings in the 16-week trial period starting from randomization visit to week 16 visit. If a participant drops out before completing the 16-week visit, all available data through the last visit date will be included for calculating CGM metrics. Minimum 168 hours of CGM data were required to calculate CGM metrics. Coefficient of Variability (CV) is the ratio of the standard deviation to the mean of the blood sugar values of each participant as measured by CGM. The reported value is the mean and standard deviation of the participant outcomes multiplied by 100. This shows the extent of the mean variability of the blood sugar values in the population. Higher CV values (up to 100) indicate greater dispersion of CGM values, which would indicate more blood sugar variability, which is considered a negative outcome. Minimum value is 0.
Time Frame: From randomization to data collection completion at the end of 16 weeks
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Closed Loop Control (CLC) | Control Group
Number analyzed (Participants) | 78 | 22
Percentage | 38 (4) | 39 (4)

9. Secondary Outcome: CGM-measured Percent of Time Above 180 mg/dL Over 12 Week Trial Extension Period
Description: Continuous Blood Glucose Monitor (CGM) values are generated every 5 minutes over the course of the study. CGM metrics were calculated by pooling all CGM readings in the 12-week period starting from the 16 week visit at the end of the main study up through the 28th week visit. If a participant drops out before completing the 28-week visit, all available data through the last visit date will be included for calculating CGM metrics. Minimum 168 hours of CGM data will be required to calculate CGM metrics. Smaller percentages of CGM-measured percentages of time above 180 mg/dL is considered a positive outcome.
Time Frame: From completion of the first 16 weeks of the main study to data collection completion at the end of 12 weeks
Measure: Mean (Standard Deviation); unit: Percentage of Time
Groups:
- Closed Loop Control (CLC) - Closed Loop Control (CLC): Eligible participants not currently using an insulin pump and Dexcom G4, G5 or Dexcom G6 CGM with minimum data requirements will initiate a run-in phase of 2 to 4 weeks that will be customized based on whether the participant is already a pump or CGM user. Participants who skip or successfully complete the run-in will be randomly assigned 3:1 to the use of closed-loop control (CLC group) system using Tandem Control-IQ Technology & Dexcom G6 CGM vs Control Group for 16 weeks. Participants randomized to the closed loop control (CLC) arm will use the t:slim X2 with Control-IQ Technology & Dexcom G6 CGM for 16 weeks. All participants will be provided the option of continue using the t:slim X2 with Control-IQ system in a 12 week Extension Phase.
  t:slim X2 with Control-IQ Technology & Dexcom G6 CGM: Eligible participants will be use the t:slim X2 with Control-IQ Technology & Dexcom G6 CGM technology for 16 weeks during the main study. All participants will be provided the option of continue using the t:slim X2 with Control-IQ system in a 12 week Extension Phase. This arm to be uset:slim X2 with Control-IQ Technology & Dexcom G6 CGM
- Control Group (SAP) - Closed Loop Control (CLC): Eligible participants not currently using an insulin pump and Dexcom G4, G5 or Dexcom G6 CGM with minimum data requirements will initiate a run-in phase of 2 to 4 weeks that will be customized based on whether the participant is already a pump or CGM user. Participants who skip or successfully complete the run-in will be randomly assigned 3:1 to the use of closed-loop control (CLC group) system using Tandem t:slim X2 with Control-IQ Technology vs Control Group for 16 weeks. All participants will be provided the option of using t:slim X2 with Control-IQ system in a 12 week Extension Phase.
  Control Group: Eligible participants will be use the study Dexcom G6 CGM for 16 weeks during the main study. All participants will be provided the option of using the t:slim X2 with Control-IQ system in a 12 week Extension Phase.
Arm/Group | Closed Loop Control (CLC) - Closed Loop Control (CLC) | Control Group (SAP) - Closed Loop Control (CLC)
Number analyzed (Participants) | 78 | 22
Percentage of Time | 33 (11) | 34 (10)

10. Secondary Outcome: CGM-measured Mean Glucose Over 12 Week Trial Extension Period
Description: Continuous Blood Glucose Monitor (CGM) values are generated every 5 minutes over the course of the study. Lower mean glucose numbers as measured by CGM in mg/dL is considered a positive outcome.
Time Frame: From completion of the first 16 weeks of the main study to data collection completion at the end of 12 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Closed Loop Control (CLC) - Closed Loop Control (CLC) | Control Group (SAP) - Closed Loop Control (CLC)
Number analyzed (Participants) | 78 | 22
mg/dL | 165 (19) | 167 (18)

11. Secondary Outcome: Glycated Hemoglobin Percent (HbA1c) at Conclusion of 12 Week Trial Extension Period
Description: Hemoglobin A1C (HbA1c) is a physiological marker of the percentage of red blood cells that have glycated (bonded with a sugar). HbA1c is used to measure changes in average blood sugar over the past three months. 5-6% is normal, 7% and above is correlated with negative long-term health outcomes.
Time Frame: At completion of the extension study, end of week 28
Measure: Mean (Standard Deviation); unit: Percent of Hemoglobin that was Glycated
Groups:
- Closed Loop Control (CLC) - Closed Loop Control (CLC): Eligible participants not currently using an insulin pump and Dexcom G4, G5 or Dexcom G6 CGM with minimum data requirements will initiate a run-in phase of 2 to 4 weeks that will be customized based on whether the participant is already a pump or CGM user. Participants who skip or successfully complete the run-in will be randomly assigned 3:1 to the use of closed-loop control (CLC group) system using Tandem Control-IQ Technology & Dexcom G6 CGM vs Control Group for 16 weeks. Participants randomized to the closed loop control (CLC) arm will use the t:slim X2 with Control-IQ Technology & Dexcom G6 CGM for 16 weeks. All participants will be provided the option of continue using the t:slim X2 with Control-IQ system in a 12 week Extension Phase.
  t:slim X2 with Control-IQ Technology & Dexcom G6 CGM: Eligible participants will be use the t:slim X2 with Control-IQ Technology & Dexcom G6 CGM technology for 16 weeks during the main study. All participants will be provided the option of continue using the t:slim X2 with Control-IQ system in a 12 week Extension Phase. This arm to be use t:slim X2 with Control-IQ Technology & Dexcom G6 CGM.
Arm/Group | Closed Loop Control (CLC) - Closed Loop Control (CLC) | Control Group (SAP) - Closed Loop Control (CLC)
Number analyzed (Participants) | 76 | 21
Percent of Hemoglobin that was Glycated | 7.2 (0.9) | 7.3 (0.7)

12. Secondary Outcome: CGM-measured Percent of Time Below 70 mg/dL Over 12 Week Trial Extension Period
Description: Continuous Blood Glucose Monitor (CGM) values are generated every 5 minutes over the course of the study. CGM measured blood sugar values below 70 mg/dL are considered to be undesirable. Thus, less time spent below 70mg/dL is considered a positive outcome.
Time Frame: From completion of the first 16 weeks of the main study to data collection completion at the end of 12 weeks
Measure: Median (Inter-Quartile Range); unit: Percentage of Time
Arm/Group | Closed Loop Control (CLC) - Closed Loop Control (CLC) | Control Group (SAP) - Closed Loop Control (CLC)
Number analyzed (Participants) | 78 | 22
Percentage of Time | 1.50 [0.64 to 2.10] | 1.34 [0.92 to 1.95]

13. Secondary Outcome: CGM-measured Percent of Time Below 54 mg/dL Over 12 Week Trial Extension Period
Description: Continuous Blood Glucose Monitor (CGM) values are generated every 5 minutes over the course of the study. CGM measured blood sugar values below 54 mg/dL have the potential to lead to unconsciousness or death. Thus, time below 54 mg/dL suggests that the person may have been close to danger.
Time Frame: From completion of the first 16 weeks of the main study to data collection completion at the end of 12 weeks
Measure: Median (Inter-Quartile Range); unit: Percentage of Time
Arm/Group | Closed Loop Control (CLC) - Closed Loop Control (CLC) | Control Group (SAP) - Closed Loop Control (CLC)
Number analyzed (Participants) | 78 | 22
Percentage of Time | 0.25 [0.09 to 0.42] | 0.25 [0.12 to 0.41]

14. Secondary Outcome: CGM-measured Percent of Time Above 250 mg/dL Over 12 Week Trial Extension Period
Description: Continuous Blood Glucose Monitor (CGM) values are generated every 5 minutes over the course of the study. CGM measured blood sugar values above 250 mg/dL are considered to be undesireable. Thus, less time spent above 250mg/dL is considered a positive outcome.
Time Frame: From completion of the first 16 weeks of the main study to data collection completion at the end of 12 weeks
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Closed Loop Control (CLC) - Closed Loop Control (CLC) | Control Group (SAP) - Closed Loop Control (CLC)
Number analyzed (Participants) | 78 | 22
percentage of time | 9.0 [6.7 to 15.4] | 10.1 [6.3 to 15.8]

15. Secondary Outcome: Continuous Glucose Monitor (CGM)-Measured Glucose Variability Percentage Measured With the Coefficient of Variation (CV) Over 12 Week Trial Extension Period
Description: Continuous Blood Glucose Monitor (CGM) values are generated every 5 minutes over the course of the study. CGM metrics were calculated by pooling all CGM readings in the 12-week trial extension period starting from 16 week visit to week 28 visit. If a participant drops out before completing the 32-week visit, all available data through the last visit date will be included for calculating CGM metrics. Minimum 168 hours of CGM data were required to calculate CGM metrics. Coefficient of Variability (CV) is the ratio of the standard deviation to the mean of the blood sugar values of each participant as measured by CGM. The reported value is the mean and standard deviation of the participant outcomes multiplied by 100. This shows the extent of the mean variability of the blood sugar values in the study group. Higher CV values (up to 100) indicate greater dispersion of CGM values, which would indicate more blood sugar variability, which is considered a negative outcome. Minimum value is 0.
Time Frame: From completion of the first 16 weeks of the main study to data collection completion at the end of 12 weeks
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Closed Loop Control (CLC) - Closed Loop Control (CLC) | Control Group (SAP) - Closed Loop Control (CLC)
Number analyzed (Participants) | 78 | 22
Percentage | 38 (4) | 38 (4)

16. Other Pre Specified Outcome: CGM-Measured Percent of Time in Range 70-140 mg/dL Over 16 Weeks
Description: Continuous Blood Glucose Monitor (CGM) values are generated every 5 minutes over the course of the study. CGM-Measured percent of time in blood sugar range 70-140 mg/dL. Larger percentages of time spent in this range is considered to be a desirable outcome.
Time Frame: From randomization to data collection completion at the end of 16 weeks
Measure: Mean (Standard Deviation); unit: Percentage of Time
Arm/Group | Closed Loop Control (CLC) | Control Group
Number analyzed (Participants) | 78 | 22
Percentage of Time | 44 (10) | 35 (11)

17. Other Pre Specified Outcome: Glucose Variability Measured With the Standard Deviation (SD) Over 16 Weeks
Description: Continuous Blood Glucose Monitor (CGM) values are generated every 5 minutes over the course of the study. CGM metrics were calculated by pooling all CGM readings in the 16-week period starting from the randomization visit up through the 16 week visit. If a participant dropped out before completing the 16-week visit, all available data through the last visit date will be included for calculating CGM metrics. Minimum 168 hours of CGM data will be required to calculate CGM metrics. Standard Deviation represents how much glucose levels fluctuate over time from a given average.
Time Frame: From randomization to data collection completion at the end of 16 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Closed Loop Control (CLC) | Control Group
Number analyzed (Participants) | 78 | 22
mg/dL | 61 (11) | 70 (13)

18. Other Pre Specified Outcome: CGM-Measured Percent of Time Below 60 mg/dL Over 16 Weeks
Description: CGM measured blood sugar values below 60 mg/dL are considered to be undesirable. Thus, less time spent below 60mg/dL is considered a positive outcome
Time Frame: From randomization to data collection completion at the end of 16 weeks
Measure: Mean (Standard Deviation); unit: Percentage of Time
Arm/Group | Closed Loop Control (CLC) | Control Group
Number analyzed (Participants) | 78 | 22
Percentage of Time | 0.67 (0.62) | 0.75 (0.55)

19. Other Pre Specified Outcome: Low Blood Glucose Index (LBGI) Over 16 Weeks
Description: Continuous Blood Glucose Monitor (CGM) metrics were calculated by pooling all CGM readings in the 16-week period starting from the randomization visit up through the 16 week visit. If a participant dropped out before completing the 16-week visit, all available data through the last visit date was included for calculating CGM metrics. Minimum 168 hours of CGM data was required to calculate CGM metrics. The low blood glucose index (LBGI) is a Glucose-variability-based metric of the risk for hypoglycemia. LBGI increases with the frequency and extent of hypoglycemic excursions and has been used as a predictor of severe events. The minimum value possible is 0, indicating no risk of low blood sugar. The maximum possible value is 100, indicating maximum possible risk of low blood sugar.
Time Frame: From randomization to data collection completion at the end of 16 weeks
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Closed Loop Control (CLC) | Control Group
Number analyzed (Participants) | 78 | 22
Score on a Scale | 0.55 (0.33) | 0.64 (0.30)

20. Other Pre Specified Outcome: Hypoglycemia Events (Defined as at Least 15 Consecutive Minutes <70 mg\dL) Over 16 Weeks
Description: A Hypoglycemic event was defined as at least 15 consecutive minutes where the CGM was lower than 70mg/dL. Fewer hypoglycemia events are considered better.
Time Frame: From randomization to data collection completion at the end of 16 weeks
Measure: Mean (Standard Deviation); unit: Hypoglycemic Event
Arm/Group | Closed Loop Control (CLC) | Control Group
Number analyzed (Participants) | 77 | 22
Hypoglycemic Event | 4.0 (2.8) | 4.6 (2.5)

21. Other Pre Specified Outcome: CGM-Measured Percent of Time >300 mg/dL Over 16 Weeks
Description: CGM measured blood sugar values above 300 mg/dL are considered to be undesirable. Thus, less time spent above 300 mg/dL is considered a positive outcome
Time Frame: From randomization to data collection completion at the end of 16 weeks
Measure: Mean (Standard Deviation); unit: Percentage of Time
Arm/Group | Closed Loop Control (CLC) | Control Group
Number analyzed (Participants) | 78 | 22
Percentage of Time | 4.1 (4.1) | 7.7 (6.3)

22. Other Pre Specified Outcome: High Blood Glucose Index (HBGI) Over 16 Weeks
Description: Continuous Blood Glucose Monitor (CGM) metrics were calculated by pooling all CGM readings in the 16-week period starting from the randomization visit up through the 16 week visit (end of study). If a participant dropped out before completing the 16-week visit, all available data through the last visit date was included for calculating CGM metrics. Minimum 168 hours of CGM data was required to calculate CGM metrics. The High Blood Glucose Index (HBGI) is a Glucose-variability-based metric of the risk for hyperglycemia that can be calculated from CGM readings. HBGI increases with the frequency and extent of hyperglycemic excursions and has been used as a predictor of severe events. The minimum value possible is 0, indicating no risk of high blood sugar. The maximum possible value is 100, indicating maximum possible risk of high blood sugar.
Time Frame: From randomization to data collection completion at the end of 16 weeks
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Closed Loop Control (CLC) | Control Group
Number analyzed (Participants) | 78 | 22
Score on a scale | 7.5 (3.1) | 10.8 (4.5)

23. Other Pre Specified Outcome: CGM-Measured Percent Time in Range 70-180 mg/dL Improvement From Baseline to 16 Weeks ≥5%
Description: This is a comparison of a binary CGM outcome indicating how many participants and what percent of participants experienced an improvement of greater than 5% in the percentage of time they were in the safe blood sugar range of 70-180 mg/dL. More participants (a greater percentage of participants) improving by this much is considered positive.
Time Frame: From randomization to data collection completion at the end of 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Closed Loop Control (CLC) | Control Group
Number analyzed (Participants) | 77 | 22
Participants | 62 | 12

24. Other Pre Specified Outcome: CGM-Measured Percent Time in Range 70-180 mg/dL Improvement From Baseline to 16 Weeks ≥10%
Description: This is a comparison of a binary CGM outcome indicating how many participants and what percent of participants experienced an improvement of greater than 10% in the percentage of time they were in the ideal blood sugar range of 70-140 mg/dL. More participants (a greater percentage of participants) improving this much is considered positive
Time Frame: From randomization to data collection completion at the end of 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Closed Loop Control (CLC) | Control Group
Number analyzed (Participants) | 77 | 22
Participants | 44 | 7

25. Other Pre Specified Outcome: Glycated Hemoglobin Percent (HbA1c) Less Than 7.0% at 16 Weeks
Description: HbA1c is a physiological marker that is used to measure changes in average blood sugar over the past three months. Numbers less than 7.0 are considered better for long-term health; thus, larger numbers or percentages of people with an HbA1c less than 7.0 is considered a positive outcome
Time Frame: From randomization to data collection completion at the end of 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Closed Loop Control (CLC) | Control Group
Number analyzed (Participants) | 77 | 22
Participants | 39 | 4

26. Other Pre Specified Outcome: Glycated Hemoglobin Percent (HbA1c) Less Than 7.5% at 16 Weeks
Description: HbA1c is a physiological marker that is used to measure changes in average blood sugar over the past three months. Numbers less than 7.5 are considered better for long-term health; thus, larger numbers or percentages of people with an HbA1c less than 7.5 is considered a positive outcome
Time Frame: From randomization to data collection completion at the end of 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Closed Loop Control (CLC) | Control Group
Number analyzed (Participants) | 77 | 22
Participants | 57 | 10

27. Other Pre Specified Outcome: Absolute Glycated Hemoglobin Percent HbA1c Improvement From Baseline to 16 Weeks Greater Than 0.5%
Description: HbA1c is a physiological marker that is used to measure changes in average blood sugar over the past three months. Improvements of 0.5% or greater are considered clinically significant improvements.
Time Frame: From randomization to data collection completion at the end of 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Closed Loop Control (CLC) | Control Group
Number analyzed (Participants) | 77 | 22
Participants | 40 | 11

28. Other Pre Specified Outcome: Absolute Glycated Hemoglobin Percent (HbA1c) Improvement From Baseline to 16 Weeks Greater Than 1.0%
Description: HbA1c is a physiological marker that is used to measure changes in average blood sugar over the past three months. Improvements of 1.0% or greater are considered clinically significant improvements
Time Frame: From randomization to data collection completion at the end of 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Closed Loop Control (CLC) | Control Group
Number analyzed (Participants) | 78 | 22
Participants | 19 | 2

29. Other Pre Specified Outcome: Glycated Hemoglobin Percent (HbA1c) Relative Improvement From Baseline to 16 Weeks Greater Than 10%
Description: as for outcome 28
Time Frame: From randomization to data collection completion at the end of 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Closed Loop Control (CLC) | Control Group
Number analyzed (Participants) | 77 | 22
Participants | 28 | 4

30. Other Pre Specified Outcome: Glycated Hemoglobin Percent HbA1c Reduction From Baseline to 16 Weeks Greater Than 1.0% or HbA1c Less Than 7.0%
Description: HbA1c is a physiological marker that is used to measure changes in average blood sugar over the past three months. Improvements of 1.0% or greater are considered clinically significant improvements, HbA1c values less than 7.0 are considered better for long-term health.
Time Frame: From randomization to data collection completion at the end of 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Closed Loop Control (CLC) | Control Group
Number analyzed (Participants) | 77 | 22
Participants | 47 | 6

31. Other Pre Specified Outcome: Fear of Hypoglycemia Survey (HFS-II) at 16 Weeks
Description: The Hypoglycemia Fear Survey-II was developed to measure behaviors and worries related to fear of hypoglycemia in adults with type 1 diabetes and was adapted for children and parents. Items are rated on a 5-point Likert scale (0=never, 4=always), with higher scores indicating higher fear of hypoglycemia. Maximum possible score: 132. Minimum possible score: 0. All questionnaires were administered online and participants/parents could skip specific questionnaires or items within a questionnaire. At least 75% of the questions must have been competed to be included in analysis. The score used for analysis was based on the average among the questions that were answered and then scaled accordingly.
Time Frame: At data collection completion at the end of 16 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Closed-Loop Control (CLC) Group (Parent Versions): Questionnaires completed by parents of participants assigned to CLC group.
- Control (SAP) Group (Parent Versions): Questionnaires completed by parents of participants assigned to Control (SAP) group.
- Closed-Loop Control (CLC) Group (Child Versions): Questionnaires completed by participants assigned to CLC group.
- Control (SAP) Group (Child Versions): Questionnaires completed by participants assigned to Control group.
Arm/Group | Closed-Loop Control (CLC) Group (Parent Versions) | Control (SAP) Group (Parent Versions) | Closed-Loop Control (CLC) Group (Child Versions) | Control (SAP) Group (Child Versions)
Number analyzed (Participants) | 78 | 22 | 78 | 22
score on a scale | 37 (13) | 45 (13) | 31 (12) | 36 (14)

32. Other Pre Specified Outcome: Clarke Hypoglycemia Awareness Scores Questionnaire at 16 Weeks
Description: The scale comprises eight questions characterizing the participant's exposure to episodes of moderate and severe hypoglycemia. It also examines the glycemic threshold for, and symptomatic responses to hypoglycemia. A score of four or more on a scale of 0 to 7 implies impaired awareness of hypoglycemia. Parents and children took the questionnaire independently.
Time Frame: At data collection completion at the end of 16 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Control (SAP) Group (Parent Versions): Questionnaires completed by parents of participants assigned to Control group.
Arm/Group | Closed-Loop Control (CLC) Group (Parent Versions) | Control (SAP) Group (Parent Versions) | Closed-Loop Control (CLC) Group (Child Versions) | Control (SAP) Group (Child Versions)
Number analyzed (Participants) | 76 | 22 | 57 | 14
score on a scale | 1.2 (1.1) | 1.6 (1.1) | 1.3 (1.1) | 1.2 (1.1)

33. Other Pre Specified Outcome: Problem Areas in Diabetes Survey (PAID) at 16 Weeks
Description: The Problem Areas In Diabetes Survey is a measure of diabetes-related emotional distress and consists of a scale of 16 items for the Parent version and 11 items for the Child version. Patients and parents rate the degree to which each item is currently problematic for them on a 6-point Likert scale, from 1 (no problem) to 6 (serious problem). Parent version maximum score: 96, minimum score 16. Child version maximum score 66, minimum score 11.
Time Frame: At data collection completion at the end of 16 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Control (SAP) Group (Child Versions): Questionnaires completed by participants assigned to Control (SAP) group.
Arm/Group | Closed-Loop Control (CLC) Group (Parent Versions) | Control (SAP) Group (Parent Versions) | Closed-Loop Control (CLC) Group (Child Versions) | Control (SAP) Group (Child Versions)
Number analyzed (Participants) | 77 | 22 | 78 | 22
units on a scale | 36 (12) | 45 (17) | 34 (16) | 37 (17)

34. Other Pre Specified Outcome: Insulin Delivery Systems: Perceptions, Ideas, Reflections and Expections (INSPIRE) Survey Scores at 16 Weeks
Description: The INSPIRE (Insulin Delivery Systems: Perceptions, Ideas, Reflections and Expectations) survey was developed to assess various aspects of a user's experience regarding automated insulin delivery for both patients and family members. The surveys include various topics important to patients with type 1 diabetes and their family members based upon >200 hours of qualitative interviews and focus groups. Response options for all surveys include a 5-point Likert scale from strongly agree to strongly disagree, along with an N/A option. Total scores on the INSPIRE questionnaires were calculated by obtaining a mean score across items, then multiplying the mean score by 25 to scale total INSPIRE measure scores from 0 to 100, with higher scores indicating greater positive expectations for automated insulin delivery systems.
Time Frame: At data collection completion at the end of 16 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Closed-Loop Control (CLC) Group (Parent Versions) | Closed-Loop Control (CLC) Group (Child Versions)
Number analyzed (Participants) | 78 | 76
score on a scale | 87 (12) | 75 (16)

35. Other Pre Specified Outcome: Pediatric Quality of Life Inventory (PedsQL Diabetes Module) at 16 Weeks
Description: This is a 33-item scale developed and validated for the measurement of diabetes-specific quality of life. Separate forms have been validated for child self-report (5-7 year old; 8-12 year old; and 12-18 year old) and parent report for these same age groups. Participants record the extent to which they (or their child) experienced each of 33 problems related to diabetes in the prior month using a 5-point Likert-type response scale (0= never a problem; 1 = almost never a problem 2 =sometimes a problem 3= often a problem 4 = almost always a problem). Items are reverse-scored and linearly transformed to a 0-100 scale (0=100, 1=7, 2=50, 3=25, 4=0) so that lower score demonstrate more diabetes symptoms and management problems, and hence lower diabetes-specific health-related quality of life. Higher scores indicate fewer symptoms or problems
Time Frame: At data collection completion at the end of 16 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Closed-Loop Control (CLC) Group (Parent Versions) | Control (SAP) Group (Parent Versions) | Closed-Loop Control (CLC) Group (Child Versions) | Control (SAP) Group (Child Versions)
Number analyzed (Participants) | 78 | 22 | 78 | 22
score on a scale | 77 (10) | 72 (12) | 76 (13) | 76 (16)

36. Other Pre Specified Outcome: Pittsburgh Sleep Quality Index (Parent Only) at 16 Weeks (Parent Only)
Description: Pittsburgh Sleep Quality Index (PSQI) is a 10-item questionnaire that measures the sleep quality and pattern of sleep in adults. Seven component scores are derived, each scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality.
Time Frame: At data collection completion at the end of 16 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Closed-Loop Control (CLC) Group (Parent Versions) | Control (SAP) Group (Parent Versions)
Number analyzed (Participants) | 73 | 20
score on a scale | 4.3 (2.9) | 6.5 (3.9)

37. Other Pre Specified Outcome: System Usability Scale (SUS) at 16 Weeks
Description: System Usability Scores (SUS)-composite score from 0 to 100 with higher scores indicating better perceived usability
Time Frame: At data collection completion at the end of 16 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Closed-Loop Control (CLC) Group (Parent Versions) | Closed-Loop Control (CLC) Group (Child Versions)
Number analyzed (Participants) | 78 | 55
score on a scale | 86 (15) | 79 (15)

38. Other Pre Specified Outcome: Total Daily Insulin (Units/kg/Day) Over 16 Weeks
Description: Total Daily Insulin (Units/kg/day) over 16 weeks. Total daily insulin dose is calculated as the sum of all insulin doses delivered by the insulin delivery system divided by the weight of the participant in kilograms and the actual duration of the treatment period in days.
Time Frame: From randomization to data collection completion at the end of 16 weeks
Measure: Mean (Standard Deviation); unit: units of insulin per kg per day
Arm/Group | Closed Loop Control (CLC) | Control Group
Number analyzed (Participants) | 78 | 21
units of insulin per kg per day | 0.94 (0.25) | 0.98 (0.32)

39. Other Pre Specified Outcome: Basal: Bolus Insulin Ratio Over 16 Weeks
Description: Insulin metrics were calculated at randomization and 16 weeks using Tandem pump data where available, otherwise using data reported on the CRF. Insulin metrics were calculated from the pump data using data in the 7 days prior to the visit. The basal:bolus ratio describes the amount of insulin used by participants to keep the blood sugar stable (basal insulin) as opposed to the amount of insulin used to metabolize consumed carbs (bolus insulin) within the total amount of insulin delivered per day.
Time Frame: 7 days leading up to the final study visit in week 16
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Closed Loop Control (CLC) | Control Group
Number analyzed (Participants) | 78 | 21
ratio | 0.87 (0.30) | 0.84 (0.38)

40. Other Pre Specified Outcome: Weight at 16 Weeks
Description: Participant Weight in kg measured at 16 weeks
Time Frame: At data collection completion at the end of 16 weeks
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Closed Loop Control (CLC) | Control Group
Number analyzed (Participants) | 78 | 21
Kg | 46 (14) | 45 (20)

41. Other Pre Specified Outcome: CGM-Measured Percent of Time in Range 70-180mg/dL Over 12 Week Trial Extension Period
Description: The primary outcome for the extension phase is improving the percent of time in the blood sugar range 70-180 mg/dL over the 12 weeks of the extension phase of the study
Time Frame: From completion of the first 16 weeks of the main study to data collection completion at the end of 12 weeks
Measure: Mean (Standard Deviation); unit: Percentage of Time
Arm/Group | Closed Loop Control (CLC) - Closed Loop Control (CLC) | Control Group (SAP) - Closed Loop Control (CLC)
Number analyzed (Participants) | 78 | 22
Percentage of Time | 66 (10) | 65 (10)

42. Other Pre Specified Outcome: CGM-Measured Percent of Time in Range 70-140 mg/dL Over 12 Week Trial Extension Period
Description: CGM-Measured percent of time in blood sugar range 70-140 mg/dL over the 12 week extension study. Larger percentages of time spent in this range is considered to be a desireable outcome.
Time Frame: From completion of the first 16 weeks of the main study to data collection completion at the end of 12 weeks
Measure: Mean (Standard Deviation); unit: Percentage of Time
Arm/Group | Closed Loop Control (CLC) - Closed Loop Control (CLC) | Control Group (SAP) - Closed Loop Control (CLC)
Number analyzed (Participants) | 78 | 22
Percentage of Time | 42 (11) | 42 (8)

43. Other Pre Specified Outcome: Glucose Variability of Blood Sugar as Measured by Continuous Glucose Monitor (CGM), Measured With the Standard Deviation (SD) Over 16 Weeks
Description: Continuous Blood Glucose Monitor (CGM) values are generated every 5 minutes over the course of the study. CGM metrics were calculated by pooling all CGM readings in the 16-week trial period starting from the randomization visit to week 16 visit. If a participant drops out before completing the 16-week visit, all available data through the last visit date will be included for calculating CGM metrics. Minimum 168 hours of CGM data were required to calculate CGM metrics. Coefficient of Variability (CV) is the ratio of the standard deviation to the mean of the blood sugar values of each participant as measured by CGM. The reported value is the mean and standard deviation of the participant outcomes multiplied by 100. This shows the extent of the mean variability of the blood sugar values in the population. Higher CV values (up to 100) indicate greater dispersion of CGM values, which would indicate more blood sugar variability, which is considered a negative outcome. Minimum value is 0.
Time Frame: From completion of the first 16 weeks of the main study to data collection completion at the end of 12 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Closed Loop Control (CLC) - Closed Loop Control (CLC) | Control Group (SAP) - Closed Loop Control (CLC)
Number analyzed (Participants) | 78 | 22
mg/dL | 62 (11) | 64 (12)

44. Other Pre Specified Outcome: Continuous Blood Glucose Monitor (CGM)-Measured Percent of Time Less Than 60 mg/dL Over 16 Weeks
Description: as for outcome 43
Time Frame: From randomization to data collection completion at the end of 16 weeks
Measure: Median (Inter-Quartile Range); unit: Percentage of Time
Arm/Group | Closed Loop Control (CLC) - Closed Loop Control (CLC) | Control Group (SAP) - Closed Loop Control (CLC)
Number analyzed (Participants) | 78 | 22
Percentage of Time | 0.48 [0.22 to 0.60] | 0.60 [0.32 to 1.19]

45. Other Pre Specified Outcome: Continuous Blood Glucose Monitor (CGM)-Measured Low Blood Glucose Index (LBGI) Over 12 Week Trial Extension Period
Description: Continuous Blood Glucose Monitor (CGM) metrics were calculated by pooling all CGM readings in the 12-week period starting from the end of the 16th week of the main trial up through the 28 week visit (end of study extension). If a participant dropped out before completing the 28-week visit, all available data through the last visit date was included for calculating CGM metrics. Minimum 168 hours of CGM data was required to calculate CGM metrics. The low blood glucose index (LBGI) is a Glucose-variability-based metric of the risk for hypoglycemia. LBGI increases with the frequency and extent of hypoglycemic excursions and has been used as a predictor of severe events. The minimum value possible is 0, indicating no risk of low blood sugar. The maximum possible value is 100, indicating maximum possible risk of low blood sugar.
Time Frame: From completion of the first 16 weeks of the main study to data collection completion at the end of 12 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Closed Loop Control (CLC) - Closed Loop Control (CLC) | Control Group (SAP) - Closed Loop Control (CLC)
Number analyzed (Participants) | 78 | 22
units on a scale | 0.48 [0.26 to 0.63] | 0.48 [0.34 to 0.58]

46. Other Pre Specified Outcome: Number of Hypoglycemia Events (Defined as at Least 15 Consecutive Minutes Less Than 70 mg\dL as Measured by Continuous Glucose Meter) Over 12 Week Trial Extension Period
Description: CGM metrics were calculated by pooling all CGM readings in the 12-week period starting from the 16th week of the main trial through the 12th week of the extension. If a participant drops out before completing the 12-week visit, all available data through the last visit date will be included for calculating CGM metrics. Minimum 168 hours of CGM data will be required to calculate CGM metrics. A hypoglycemic event is defined as 15 consecutive minutes with a sensor glucose value below 54 mg/dL. Fewer glycemic events per week is considered a better outcome.
Time Frame: From completion of the first 16 weeks of the main study to data collection completion at the end of 12 weeks
Measure: Median (Inter-Quartile Range); unit: Hypoglycemic Event
Arm/Group | Closed Loop Control (CLC) - Closed Loop Control (CLC) | Control Group (SAP) - Closed Loop Control (CLC)
Number analyzed (Participants) | 78 | 22
Hypoglycemic Event | 3.4 [1.4 to 5.2] | 2.9 [2.8 to 4.1]

47. Other Pre Specified Outcome: CGM-Measured Percent of Time Above 300 mg/dL Over 12 Week Trial Extension Period
Description: CGM measured blood sugar values above 300 mg/dL are considered to be undesireable. Thus, less time spent above 300mg/dL is considered a positive outcome
Time Frame: From completion of the first 16 weeks of the main study to data collection completion at the end of 12 weeks
Measure: Median (Inter-Quartile Range); unit: Percentage of Time
Arm/Group | Closed Loop Control (CLC) - Closed Loop Control (CLC) | Control Group (SAP) - Closed Loop Control (CLC)
Number analyzed (Participants) | 78 | 22
Percentage of Time | 2.9 [1.8 to 5.9] | 3.5 [1.8 to 6.6]

48. Other Pre Specified Outcome: High Blood Glucose Index (HBGI) Over 12 Weeks of Trial Extension Period
Description: Continuous Blood Glucose Monitor (CGM) metrics were calculated by pooling all CGM readings in the 12-week period starting from the end of the 16th week of the main trial up through the 28 week visit (end of study extension). If a participant dropped out before completing the 28-week visit, all available data through the last visit date was included for calculating CGM metrics. Minimum 168 hours of CGM data was required to calculate CGM metrics. The High Blood Glucose Index (HBGI) is a Glucose-variability-based metric of the risk for hyperglycemia that can be calculated from CGM readings. HBGI increases with the frequency and extent of hyperglycemic excursions and has been used as a predictor of severe events. The minimum value possible is 0, indicating no risk of high blood sugar. The maximum possible value is 100, indicating maximum possible risk of high blood sugar.
Time Frame: From completion of the first 16 weeks of the main study to data collection completion at the end of 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Closed Loop Control (CLC) - Closed Loop Control (CLC) | Control Group (SAP) - Closed Loop Control (CLC)
Number analyzed (Participants) | 78 | 22
units on a scale | 8.0 (3.3) | 8.3 (3.2)

49. Other Pre Specified Outcome: Glycated Hemoglobin Percent (HbA1c) Less Than 7.0% at Conclusion of 12 Week Trial Extension Period
Description: as for outcome 25
Time Frame: At completion of the extension study, end of week 28
Measure: Count of Participants; unit: Participants
Arm/Group | Closed Loop Control (CLC) - Closed Loop Control (CLC) | Control Group (SAP) - Closed Loop Control (CLC)
Number analyzed (Participants) | 76 | 21
Participants | 32 | 4

50. Other Pre Specified Outcome: Glycated Hemoglobin Percent (HbA1c) Less Than 7.5% at Conclusion of 12 Week Trial Extension Period
Description: as for outcome 26
Time Frame: At completion of the extension study, end of week 28
Measure: Count of Participants; unit: Participants
Arm/Group | Closed Loop Control (CLC) - Closed Loop Control (CLC) | Control Group (SAP) - Closed Loop Control (CLC)
Number analyzed (Participants) | 76 | 21
Participants | 48 | 13

51. Other Pre Specified Outcome: Fear of Hypoglycemia Survey (HFS-II) at Conclusion of 12 Week Trial Extension Period
Description: as for outcome 31
Time Frame: At completion of the extension study, end of week 28
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- CLC-CLC Group (Parent Versions): Questionnaires completed by parents of participants assigned to CLC-CLC group.
- SAP-CLC Group (Parent Versions): Questionnaires completed by parents of participants assigned to SAP-CLC group.
- CLC-CLC Group (Child Versions): Questionnaires completed by participants assigned to CLC-CLC group.
- SAP-CLC Group (Child Versions): Questionnaires completed by participants assigned to SAP-CLC group.
Arm/Group | CLC-CLC Group (Parent Versions) | SAP-CLC Group (Parent Versions) | CLC-CLC Group (Child Versions) | SAP-CLC Group (Child Versions)
Number analyzed (Participants) | 78 | 22 | 78 | 22
score on a scale | 36 (12) | 43 (17) | 30 (11) | 32 (14)

52. Other Pre Specified Outcome: Clarke Hypoglycemia Awareness Scores Questionnaire at Conclusion of 12 Week Trial Extension Period
Description: The scale comprises eight questions characterizing the participant's exposure to episodes of moderate and severe hypoglycemia. It also examines the glycemic threshold for, and symptomatic responses to hypoglycemia. A score of four or more on a scale of 0 to 7 implies impaired awareness of hypoglycemia.
Time Frame: At completion of the extension study, end of week 28
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CLC-CLC Group (Parent Versions) | SAP-CLC Group (Parent Versions) | CLC-CLC Group (Child Versions) | SAP-CLC Group (Child Versions)
Number analyzed (Participants) | 78 | 21 | 57 | 14
score on a scale | 1.1 (1.1) | 1.5 (1.2) | 1.5 (1.2) | 1.7 (1.1)

53. Other Pre Specified Outcome: Problem Areas in Diabetes Survey (PAID) at Conclusion of 12 Week Trial Extension Period
Description: as for outcome 33
Time Frame: At completion of the extension study, end of week 28
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CLC-CLC Group (Parent Versions) | SAP-CLC Group (Parent Versions) | CLC-CLC Group (Child Versions) | SAP-CLC Group (Child Versions)
Number analyzed (Participants) | 78 | 22 | 78 | 22
score on a scale | 36 (13) | 40 (17) | 30 (11) | 37 (19)

54. Other Pre Specified Outcome: Insulin Delivery Systems: Perceptions, Ideas, Reflections and Expectations (INSPIRE) Survey Scores at Conclusion of 12 Week Trial Extension Period
Description: as for outcome 34
Time Frame: At completion of the extension study, end of week 28
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CLC-CLC Group (Parent Versions) | SAP-CLC Group (Parent Versions) | CLC-CLC Group (Child Versions) | SAP-CLC Group (Child Versions)
Number analyzed (Participants) | 78 | 22 | 77 | 22
score on a scale | 89 (12) | 86 (17) | 76 (17) | 78 (14)

55. Other Pre Specified Outcome: Pediatric Quality of Life Inventory (PedsQL Diabetes Module) at Conclusion of 12 Week Trial Extension Period
Description: as for outcome 35
Time Frame: At completion of the extension study, end of week 28
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CLC-CLC Group (Parent Versions) | SAP-CLC Group (Parent Versions) | CLC-CLC Group (Child Versions) | SAP-CLC Group (Child Versions)
Number analyzed (Participants) | 78 | 22 | 78 | 22
score on a scale | 77 (11) | 77 (15) | 78 (13) | 77 (18)

56. Other Pre Specified Outcome: Pittsburgh Sleep Quality Index (Parent Only) at Conclusion of 12 Week Trial Extension Period
Description: as for outcome 36
Time Frame: At completion of the extension study, end of week 28
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CLC-CLC Group (Parent Versions) | SAP-CLC Group (Parent Versions)
Number analyzed (Participants) | 74 | 20
score on a scale | 4.4 (2.9) | 5.4 (3.6)

57. Other Pre Specified Outcome: System Usability Scale (SUS) at Conclusion of 12 Week Trial Extension Period
Description: System Usability Scores (SUS)-composite score from 0 to 100 with higher scores indicating better perceived usability.
Time Frame: At completion of the extension study, end of week 28
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CLC-CLC Group (Parent Versions) | SAP-CLC Group (Parent Versions) | CLC-CLC Group (Child Versions) | SAP-CLC Group (Child Versions)
Number analyzed (Participants) | 77 | 22 | 56 | 14
score on a scale | 86 (21) | 84 (22) | 81 (18) | 83 (10)

58. Other Pre Specified Outcome: Total Daily Insulin (TDI) (Units/kg/Day) Over 12 Week Trial Extension Period
Description: Total Daily Insulin (Units/kg/day) over 12 weeks. Total daily insulin dose is calculated as the sum of all insulin doses delivered by the insulin delivery system divided by the weight of the participant in kilograms and the actual duration of the treatment period in days.
Time Frame: From completion of the first 16 weeks of the main study to data collection completion at the end of 12 weeks
Measure: Mean (Standard Deviation); unit: units of insulin per kg per day
Arm/Group | Closed Loop Control (CLC) - Closed Loop Control (CLC) | Control Group (SAP) - Closed Loop Control (CLC)
Number analyzed (Participants) | 76 | 22
units of insulin per kg per day | 0.93 (0.25) | 1.04 (0.34)

59. Other Pre Specified Outcome: Basal: Bolus Insulin Ratio at Conclusion of 12 Week Trial Extension Period
Description: Insulin metrics were calculated at 16 weeks and 28 weeks using Tandem pump data where available, otherwise using data reported on the CRF. Insulin metrics were calculated from the pump data using data in the 7 days prior to the visit. The basal:bolus ratio describes the amount of insulin used by participants to keep the blood sugar stable (basal insulin) as opposed to the amount of insulin used to metabolize consumed carbs (bolus insulin) within the total amount of insulin delivered per day.
Time Frame: 7 days leading up to the final extension study visit in week 28
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Closed Loop Control (CLC) - Closed Loop Control (CLC) | Control Group (SAP) - Closed Loop Control (CLC)
Number analyzed (Participants) | 76 | 22
ratio | 0.84 [0.71 to 1.10] | 1.0 [0.83 to 1.47]

60. Other Pre Specified Outcome: Body Mass Index (BMI) at Conclusion of 12 Week Trial Extension Period
Description: Body Mass Index (BMI) is a calculation of participant body weight in kilograms and height in centimeters. The z-score was calculated from values taken at the end of the 28 weeks of the study. Z-score of zero represents the US population mean for their age and sex group. Positive Z scores indicate higher body mass index values than the population mean, which is generally considered undesirable
Time Frame: At completion of the extension study, end of week 28
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Closed Loop Control (CLC) - Closed Loop Control (CLC) | Control Group (SAP) - Closed Loop Control (CLC)
Number analyzed (Participants) | 76 | 22
Z-score | .46 (0.97) | 0.68 (1.03)

ADVERSE EVENTS:
Time Frame: 28 weeks
Groups:
- Closed Loop Control up to 16 Weeks (Main Study): Eligible participants not currently using an insulin pump and Dexcom G4, G5 or Dexcom G6 CGM with minimum data requirements initiated a run-in phase of 2 to 4 weeks that was customized based on whether the participant is already a pump or CGM user. Participants who skipped or successfully completed the run-in were randomly assigned 3:1 to the use of closed-loop control (CLC group) system using Tandem Control-IQ Technology & Dexcom G6 CGM vs Control Group for 16 weeks. Participants randomized to the closed loop control (CLC) arm used the t:slim X2 with Control-IQ Technology & Dexcom G6 CGM for 16 weeks.
- Standard of Care up to 16 Weeks (Main Study): Eligible participants not currently using an insulin pump and Dexcom G4, G5 or Dexcom G6 CGM with minimum data requirements initiated a run-in phase of 2 to 4 weeks that was customized based on whether the participant is already a pump or CGM user. Participants who skipped or successfully completed the run-in were randomly assigned 3:1 to the use of closed-loop control (CLC group) system using Tandem t:slim X2 with Control-IQ Technology vs Control Group for 16 weeks.
- Continued Closed Loop Control Week 16 to Week 28 (Extension Study); Standard of Care to Closed Loop Control Week 16 to Week 28 (Extension Study): All participants were provided the option of continuing to use the t:slim X2 & Dexcom G6 CGM technology with Control-IQ system in a 12 week Extension Phase.
Arm/Group | Closed Loop Control up to 16 Weeks (Main Study) | Standard of Care up to 16 Weeks (Main Study) | Continued Closed Loop Control Week 16 to Week 28 (Extension Study) | Standard of Care to Closed Loop Control Week 16 to Week 28 (Extension Study)
All-Cause Mortality (participants affected / at risk) | 0/78 | 0/23 | 0/78 | 0/22
Serious Adverse Events (participants affected / at risk) | 1/78 | 0/23 | 0/78 | 0/22
Other Adverse Events (participants affected / at risk) | 15/78 | 2/23 | 6/78 | 2/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Closed Loop Control up to 16 Weeks (Main Study) (N=78) | Standard of Care up to 16 Weeks (Main Study) (N=23) | Continued Closed Loop Control Week 16 to Week 28 (Extension Study) (N=78) | Standard of Care to Closed Loop Control Week 16 to Week 28 (Extension Study) (N=22)
Hospitalization for Gastroenteritis Leading to Ketosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — The serious adverse event was hospitalization for gastroenteritis leading to ketosis, which was determined not to be related to trial device, as assessed by a trial investigator and adjudicated by the medical monitor.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Closed Loop Control up to 16 Weeks (Main Study) (N=78) | Standard of Care up to 16 Weeks (Main Study) (N=23) | Continued Closed Loop Control Week 16 to Week 28 (Extension Study) (N=78) | Standard of Care to Closed Loop Control Week 16 to Week 28 (Extension Study) (N=22)
Abscess at sensor site (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hyperglycemia (Endocrine disorders) | 2 (2) | 0 (0) | 6 (7) | 1 (2)
Ketosis (Endocrine disorders) | 12 (12) | 1 (1) | 0 (0) | 1 (1)
Accidental over-delivery of insulin (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoglycemia (Endocrine disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Baseline Measures Overview - Missing data (CLC/SAP): annual household income 4 (5%)/2 (9%), TDI 1 (1%)/0 (0%). Very little missing CGM data: one participant was missing baseline data; another participant was missing follow-up data. Both participants were included in the model for the timepoint with available data so each had one record in the dataset instead of two. This direct likelihood method therefore maximizes the likelihood function integrated over possible values of the missing data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2019-10-09): https://cdn.clinicaltrials.gov/large-docs/89/NCT03844789/Prot_001.pdf
  • Statistical Analysis Plan (2019-12-20): https://cdn.clinicaltrials.gov/large-docs/89/NCT03844789/SAP_002.pdf
  • Informed Consent Form (2019-01-25): https://cdn.clinicaltrials.gov/large-docs/89/NCT03844789/ICF_000.pdf